CLINICAL TRIAL: NCT01376544
Title: Randomised Trial Comparing Assist Control Ventilation to Pressure Support Ventilation During Weaning
Brief Title: Trial of Weaning by Synchronized Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Professor Anne Greenough, King's College London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07/H0808/147
Record Dates: First submitted 2011-05-26; First posted 2011-06-20 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-06

CONDITIONS: Neonatal Respiratory Failure
Keywords: Neonate; Weaning; Assist control ventilation; Pressure support ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Assist control ventilation (Active Comparator): Assist control ventilation
  Interventions: Device: Treatment protocol designed to evaluate (SLE 5000 ventilator)
- Pressure support ventilation (Active Comparator)
  Interventions: Device: Treatment protocol designed to evaluate (SLE 5000 ventilator)

INTERVENTIONS:
Device: Treatment protocol designed to evaluate (SLE 5000 ventilator) — Assist control ventilation and pressure support ventilation
  Other Names: SLE 5000 ventilator

SUMMARY:
During assist control ventilation and pressure support ventilation (PSV), the start of ventilator inflation is determined by the start of the infant's inspiratory effort. During PSV, termination of inflation is determined by the level of the infant's inspiratory flow. In a randomized trial, no significant differences were found between assist control and pressure support ventilation with regard to the duration of weaning, time to successful extubation, work of breathing, rate of asynchrony and level of respiratory muscle strength.

DETAILED DESCRIPTION:
Objectives: To test the hypothesis that the duration of weaning would be shorter using assist control ventilation (ACV) rather than pressure support ventilation (PSV). To determine if any differences in the duration of weaning reflected differences in the work of breathing, the rate of asynchrony or the level of respiratory muscle strength.

Patients and methods: Thirty-six infants, median gestational age 29 (range 24 to 39) weeks, were randomized to weaning by either ACV or PSV. The duration of weaning was recorded. At baseline (study entry), 24 hours after entering the study and immediately prior to extubation, the work of breathing was assessed by measuring the transdiaphragmatic pressure time product (PTPdi), thoracoabdominal asynchrony (TAA) was assessed using respiratory inductance plethysmography and respiratory muscle strength measured by recording the maximal inspiratory pressure produced during an airway occlusion during crying (Pimax). Immediately prior to extubation, the level of active expiration was also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Ventilated neonates less than 14 days of age

Exclusion Criteria:

* Congenital heart disease, hypoxic ischaemic encephalopathy

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2008-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To determine which mode of ventilation was associated with a shorter duration of weaning. | Up to 28 days after birth

SECONDARY OUTCOMES:
Change in Work of breathing thoraco-abdominal asynchrony respiratory muscle strength | Baseline, 24 hours and prior to extubation

CONTACTS AND LOCATIONS:
Overall Officials: Anne Greenough, MD, Principal Investigator — King's College London
Locations (1):
- Neonatal Intensive Care Unit, London, United Kingdom